CLINICAL TRIAL: NCT00692744
Title: Study of Quality of Life After Aneurysmal Subarachnoid Hemorrhage in Patients Aged 70 Years or Older.
Brief Title: Quality of Life in Elderly After Aneurysmal Subarachnoid Hemorrhage (SAH)
Acronym: FASHE
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/042/HP
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Hydrocephalus; Cerebral Vasospasm
Keywords: Subarachnoid hemorrhage; Cerebral aneurysm; Elderly
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hydrocephalus; Vasospasm, Intracranial; Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 2 randomized arms (clipping and coiling) and 3 prospective observational arms (clipping, coiling, conservative) For the randomized arms, we anticipated 20 patients in each arm.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Randomized microsurgical: After randomization, this group was constituted of patients treated by microsurgical clipping.
- Randomized endovascular: After randomization, this group was constituted of patients treated by endovascular coiling.
- Prospective observational microsurgical: The randomization was ethically unsuitable because of the aneurysm predisposed to the microsurgical clipping after discussion into the neurovascular interdisciplinary team.
- Prospective observational endovascular: The randomization was ethically unsuitable because of the aneurysm morphology predisposed to the endovascular coiling after discussion into the neurovascular interdisciplinary team.
- Prospective observational conservative: This group was constituted of patients whom no curative treatment of the aneurysm sac could not be proposed.

SUMMARY:
In all the Western populations, the annual incidence of subarachnoid hemorrhage (SAH) increase with age. In patients older than 70 years, the occurrence of SAH exposes them to high risk of morbidity and a poor quality of life.

In this age bracket, the single randomized which compared endovascular coiling to microsurgical clipping (ISAT Study) showed that the relative risk of morbidity increased after coiling. Moreover, some prospectives studies about endovascular coiling described favorable outcome in 48% to 63% of patients, complete occlusion in 51% to 69% and a procedural complication rate in 13% to 19%. From prospectives series, the proportion of favorable outcome after microsurgical clipping was estimated around 66% but the procedural complications are few reported. The outcome for patients treated conservatively was catastrophic. Lastly, the hydrocephalus in this age class is common, occurring in 55% of patients.

The study hypothesis is that, in this age class, no difference exists between the 2 obliteration procedures.

An accurate evaluation of result in term of functional disability, quality of life and prognosis predictive factors seems a judicious question.

DETAILED DESCRIPTION:
The aim of our study was to determine a significant difference in terms of functional disability between microsurgical clipping and endovascular coiling in the elderly population.

Randomized multicenter trial: 2 randomized arms (clipping and coiling) plus 3 observational prospective arms (clipping, coiling, conservative).

Inclusion time: 48 months. Follow up: 12 months. Monitoring: 6 months. Duration of the trial: 66 months. Major end point: proportion of patients with unfavourable outcome at 12 months (mRS > 2).

Secondary end point: Quality of life at 12 months (EORTC scale), causes of morbidity (mRS > 2) and mortality, Dysautonomia according to the ADL and IADL scales.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old and more
* Subarachnoid hemorrhage in grade I-IV of WFNS scale
* Ruptured cerebral aneurysm diagnosed on multislice computed tomography angiography or cerebral angiography
* treatment of subarachnoid hemorrhage

Exclusion Criteria:

* Patients in grade V of WFNS scale
* Subarachnoid hemorrhage without cerebral aneurysm
* Patients with cerebral dementia, neurologic or psychiatric antecedents

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Primary cara clinic in differents countries of France
Sampling Method: Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2008-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 12 months

SECONDARY OUTCOMES:
Min Mental State Examination | 12 months
Quality of LIfe, QLQ C30 questionnaire from EORTC | 12 months
Self-maintaining and instrumental activities of daily living, ADL and IADL score | 12 months
Hydrocephalus and risk factors | 12 months
Causes of morbidity and mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: François PROUST, M.D., Ph.D., Principal Investigator — University Hospital, Rouen; Serge BRACARD, M.D., Ph.D., Principal Investigator — Central Hospital, Nancy, France; Guillaume PENCHET, M.D., Study Director — University Hospital, Bordeaux; Evelyne EMERY, M.D., Study Director — University Hospital, Caen; Bernard IRTHUM, M.D., Study Director — Clermont University Hospital; Klaus MOURIER, M.D., Study Director — Centre Hospitalier Universitaire Dijon; Emmanuel GAY, M.D., Study Director — University Hospital, Grenoble; Jean-Paul LEJEUNE, M.D., Study Director — Lille University Hospital; Isabelle PELISSOU, M.D., Study Director — Hospices Civils de Lyon; Pierre Hughes ROCHE, M.D., Study Director — University Hospital, Marseille; Thierry CIVIT, M.D., Study Director — Central Hospital, Nancy, France; Michel LONJON, M.D., Study Director — Nice University Hospital; Philippe DAVID, M.D., Study Director — Paris University Hospital; Benoit BATAILLE, M.D., Study Director — Poitiers University Hospital; Xavier MORANDI, M.D., Study Director — Rennes University Hospital; Jacques LAGUARRIGUE, M.D., Study Director — University Hospital, Toulouse; Romain BILLON-GRAND, M.D., Study Director — Besançon University Hospital; Damien BRESSON, M.D., Study Director — Paris University Hospital
Locations (2):
- France (2):
  - PROUST, Rouen
  - Rouen University Hospital, Rouen

REFERENCES:
- [Background] Proust F, Gerardin E, Derrey S, Lesveque S, Ramos S, Langlois O, Tollard E, Benichou J, Chassagne P, Clavier E, Freger P. Interdisciplinary treatment of ruptured cerebral aneurysms in elderly patients. J Neurosurg. 2010 Jun;112(6):1200-7. doi: 10.3171/2009.10.JNS08754. PMID 19961311
- [Background] Proust F, Bracard S, Thines L, Leclerc X, Penchet G, Berge J, Vignes JR, Irthum B, Gabrillargues J, Chazal J, Bataille B, Drouinau J, Mourier K, Ricolfi F, Gay E, Bessou P, Lonjon M, Sedat J, David P, Lajaunias P, Morandi X, Gauvrit JY, Pelissou I, Turjman F, Roche PH, Dufour H, Levrier O, Emery E, Courtheoux P, Laguarrigue J, Cognard C, Civit T, Lejeune JP. [Aneurismal subarachnoid hemorrhage in the elderly subject. Should this patient participate in a randomized clinical trial?]. Neurochirurgie. 2010 Feb;56(1):67-72. doi: 10.1016/j.neuchi.2009.11.002. Epub 2010 Jan 8. No abstract available. French. PMID 20060549